CLINICAL TRIAL: NCT06445907
Title: Phase I Study of Q702 With Azacitidine and Venetoclax for Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0178; NCI-2024-04788 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Dose Escalation) (Experimental): Participants receive Q702 orally (PO) once daily (QD) on days 1-7 and 15-21 of each cycle. Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7 of each cycle and venetoclax PO QD on days 1-21 or days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also undergo collection of blood samples and bone marrow aspiration and/or biopsy throughout the trial.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Q702
- Part 2 (Dose Expansion) (Experimental): Participants receive Q702 orally (PO) once daily (QD) on days 1-7 and 15-21 of each cycle. Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7 of each cycle and venetoclax PO QD on days 1-21 or days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also undergo collection of blood samples and bone marrow aspiration and/or biopsy throughout the trial.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Q702

INTERVENTIONS:
Drug: Azacitidine — Given by IV
  Other Names: 5-azacytidine; 5-aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Q702 — Given by PO

SUMMARY:
To learn about the safety and tolerability of the drug combination of Q702, azacitidine, and venetoclax when given to participants with relapsed/refractory AML.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate safety of Q702 and the combination of azacitidine, venetoclax.

Secondary Objectives:

* To estimate rate of CR/CRh/CRi by 4 treatment cycles
* To estimate overall response rate (ORR)
* To estimate rate of MRD negative by 4 treatment cycles
* To estimate overall survival (OS)
* To estimate relapse-free survival (RFS)

Exploratory Objectives:

* To determine the plasma concentration and pharmacokinetic (PK) parameters of Q702 when dosed in combination with azole antifungals in AML patients
* To estimate duration of response (DOR)
* To estimate median time to blood count recovery
* To estimate median time to first response
* To estimate median time to negative MRD
* To study drug-drug interactions with CYP3A4 inhibitor azole antifungals
* Additional response and survival endpoints
* To explore biomarkers of response, pathway engagement, and resistance

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to have a confirmed diagnosis of AML, or MDS/AML with 10% to 19% blasts, per the International Consensus Classification 2022 or the WHO 2022 classification.23,24
2. Patients .18 years with R/R AML or R/R MDS/AML, other than acute promyelocytic leukemia (APL), with no available standard treatment options.
3. Relapsed or refractory disease defined by standard criteria as follows:

   a. Relapsed: Bone marrow blasts .5%, reappearance of blasts in the blood, or development of extramedullary disease following achievement of CR/CRi/MLFS b. Refractory: Failure to achieve CR/CRi/MLFS following initial treatment, with evidence of persistent leukemia by blood and/or bone marrow evaluation with blasts .5% c. Appropriate prior therapy in order for patient to be deemed relapsed or refractory include any of the following: i. At least 1 cycle of purine analogue containing intensive induction chemotherapy regimen, e.g., FLAG-Ida, CLIA or CLAG-M or similar regimens with or without venetoclax.25,26 ii. At least 1 cycle of intensive induction chemotherapy with venetoclax, e.g., 7 + 3 or CPX-351 with venetoclax or similar regimens iii. At least 2 cycles of intensive induction chemotherapy such as 7 + 3 or 5 + 2 or similar regimens without venetoclax iv. 2 cycles of BCL2 inhibitor with HMA/LDAC +/- other agents v. 4 cycles of HMA-based regimen without BCL2 inhibitor

   - Younger/fit patients (<60 years) in first relapse following intensive chemotherapy, will only be eligible if the first remission (CR1) duration was .12 months.

   d. Patients relapsing with persistent or new TP53 mutation will be eligible irrespective of CR1 duration. e. Older/unfit patients who relapse on HMA + venetoclax based maintenance regimen will be eligible irrespective of CR1 duration.
4. ECOG PS 0 to 1
5. Patients relapsing after allo-SCT may be eligible if they have recovered from all transplant related toxicities and are off all immunosuppression, with no more than grade 1 chronic GVHD. Physiologic ( greplacement h) dose of steroids (.10 mg prednisone or equivalent) may be acceptable. Patients must be off all immunosuppression, including calcineurin inhibitors, for at least 2 weeks or 5 half-lives, whichever is longer, prior to enrollment on study.
6. Patients with actionable mutations with available FDA-approved therapies, e.g., FLT3, IDH1/2 inhibitors may be enrolled after they have exhausted appropriate lines of FDA approved treatment options.
7. Patients with antecedent hematological disorder (AHD), e.g., aplastic anemia, myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML) or myeloproliferative disorder or neoplasm (MPD or MPN) who have previously received a regimen appropriate for AML for the antecedent hematological disorder, as described above, and have progressed to AML, will be eligible for the dose escalation and salvage dose expansion cohorts. This is due to recognized poor outcomes in such patients with "treated secondary AML".27,28
8. Adequate hepatic function (total bilirubin . 1.5 x upper limit of normal (ULN), and AST and/or ALT . 2 x ULN). Patients with Gilbert disease will be eligible with total bilirubin . 4.5 mg/dL.
9. Adequate renal function with creatinine clearance . 60 mL/min calculated by the Cockcroft- Gault formula or MDRD equation or measured by 24-hour urine collection.
10. The effects of these agents on the developing human fetus are unknown. For this reason, and because other therapeutic agents used in this trial may be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 90 days after last treatment.

    a. This includes all female patients between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: i. Postmenopausal (no menses in greater than or equal to 12 consecutive months).

    ii. History of hysterectomy or bilateral salpingo-oophorectomy. iii. Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range, who have received whole pelvic radiation therapy).

    iv. History of bilateral tubal ligation or another surgical sterilization procedure.

    b. Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    c. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with t(15;17) karyotypic abnormality.
2. Patient has a white blood cell count > 15 x 10./L. Hydroxyurea, and/or cytarabine (up to 2 g/m2 total) used as supportive care is permitted to meet this criterion prior to enrollment.
3. Prior use of any cytotoxic chemotherapy, targeted therapy, radiation therapy, immunotherapy, or other clinical trial therapies within 2 weeks or 5 half-lives, whichever is shorter, prior to first dose of study treatment. Patients should have recovered from all prior therapy related toxicities. Patients may receive hydroxyurea or cytarabine for control of WBC count during this washout period.
4. Patients with known symptomatic or uncontrolled CNS leukemia.
5. Patient has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
6. Active ophthalmological disorders, e.g., retinal pigment epithelium (RPE)/photoreceptor disorders such as retinitis pigmentosa, cone-rod dystrophies, Bests dystrophy, Stargardt disease (STGD), macular degeneration. Exceptions:

   1. Mild blurry vision, either age-related or due to ocular or systemic disorder (e.g., diabetes, dry eyes, cataracts, uncorrected refraction abnormality) may be allowed at the discretion of an ophthalmologist if deemed as not constituting evidence of preexisting retinopathy or a condition with the potential to cause a predisposition to druginduced retinopathy.
   2. Patients with only one assessable eye and no evidence of pre-existing retinopathy may be allowed at the discretion of the principal investigator.
7. Any known and active neurological disorder with residual neurological deficit or requiring pharmacotherapy.
8. Patients with known acute or chronic liver disease, cirrhosis, hepatic steatosis with elevated liver function tests or elevated LFTs of unknown etiology.
9. Active and uncontrolled comorbidities including decompensated congestive heart failure NYHA class III/IV, clinically significant, uncontrolled arrhythmia, acute respiratory failure, unstable or decompensated pulmonary disease, as judged by the treating physician.
10. Decompensated congestive heart failure, hypokalemia, prolonged QT interval corrected for heart rate (QTc) to greater than 470 msec or long QT syndrome, or history of Torsades de pointes. Appropriate corrections may be applied for patients with bundle branch block.
11. Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications as determined by the investigator.
12. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection with detectable viral DNA or RNA, respectively, or known HIV or HTLV-1 infection.
13. Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator.
14. Any previous malignancy, except when the patient has completed definitive curative-intent treatment with chemotherapy and/or surgery and/or radiotherapy at least 1 month prior to enrollment. Patients having completed definitive treatment for the following conditions may be eligible immediately after completion of definitive curative-intent therapy, after healing of wounds, and no evidence of residual disease by examination or imaging or cytology/pathology, e.g., non-melanoma skin cancers, or any carcinoma in-situ, e.g., ductal carcinoma in situ, urothelial cancer, cervical cancer, localized prostate cancer, pre-cancerous colon polyp, etc.
15. Major surgery within 4 weeks prior to screening or a major wound that has not fully healed.
16. Patients under legal protection measure (guardianship, trusteeship or safeguard of justice) and/or uncontrolled psychiatric comorbidities, ongoing illicit substance abuse, any impairment or unwillingness to comply with the treatments, follow-up, requirements and procedures of this clinical trial.
17. A known hypersensitivity or severe allergy to study drug components or diluents
18. Nursing women, women of childbearing potential (WOCBP) with positive urine or serum pregnancy test, or WOCBP who are not willing to maintain adequate contraception.
19. Pregnant women are excluded from this study because study agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (Aes) in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org